CLINICAL TRIAL: NCT01141023
Title: The Parkinson's Progression Markers Initiative (PPMI)
Brief Title: Study to Identify Clinical, Imaging and Biologic Markers of Parkinson Disease Progression
Acronym: PPMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ken Marek, MD (Other)
Collaborators: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor-Investigator, Ken Marek, MD, Study Chair, Michael J. Fox Foundation for Parkinson's Research
Organization: Michael J. Fox Foundation for Parkinson's Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PPMI-001
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Bio-markers; Neurodegenerative disorder; Imaging; Prodromal
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — ioflupane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Datscan SPECT Imaging (Experimental): Subjects will b injected with 3-5 mCi of dopamine transporter. Within a 4 hour (+/- 30 minutes) window following the injection, subjects will undergo SPECT imaging on the camera.
  Interventions: Drug: DaTscan

INTERVENTIONS:
Drug: DaTscan
  Other Names: Ioflupane

SUMMARY:
This is a observational, multi-center study to assess progression of clinical features, imaging and biologic biomarkers in Parkinson disease (PD) patients compared to healthy controls (HC) and in PD patient subtypes.

The primary objective of this study is to identify clinical, imaging and biologic markers of PD progression for use in clinical trials of disease-modifying therapies.

DETAILED DESCRIPTION:
Amendment 14 - 26-Mar-2018 Revised to reflect the implementation of PPMI Wearables and Sensor Study Companion Protocol

Amendment 13 - 20-Nov-2017 Extension of study duration until 2023 for all cohorts (except Genetic Registry).

Amendment 12 - 01-Jun-2017 Planned date of trial extended to September 30, 2020 Ceasing new enrollments into the Genetic Registry for LRRK2 and GBA subjects Added Sensor - PPMI Companion Study Allow for consent to share contact information with FOUND team at any visit. Incorporation of Parkinson's Disease Risk Factor Questionnaire (PD-RFQ) into FOUND.

Amendment 11 - 01-Apr-2016 Added the collection of peripheral blood mononuclear cells (PBMC) from blood samples at interim visits.

Addition of PPMI Pathology Core/PPMI Brain and Tissue Bank Addition of Gait Assessment Companion Study (Select PPMI sites - Genetic Cohort only) Testing for additional GBA mutations - previously testing involved testing only for the GBA N370S mutation; however, going forward, testing will include tests for additional GBA mutations that are identified as being associated with certain ancestry.

Amendment 10 - 05-Oct-2015 Extended study period for PD and Healthy Control subjects through 8 years. For Prodromal subjects (RBD and Hyposmic) added iPSC companion study.

Amendment 9 - 01-Nov-2014 Addition of GBA throughout to document additional testing for GBA mutation. Allocation of subjects in Genetic Cohort and Genetic Registry revised to account for inclusion of GBA subjects.

Amendment 8 - 12-May-2014 Companion Protocols: skin biopsy/stem cell; Amyloid Imaging 18F Florbetaben; Family History Sub-Study; FOUND in PPMI registry. More detailed description of new procedures including: Advance directive for clinical research participation; Extension of study period (for SWEDDs with positive scans at Yr. 2) by continuing or re-inviting to study and followed (as per PD subjects through Month 60); Objective Parkinson Disease Measurement (OPDM) finger tapping measurement.

Amendment 7 - 14-Oct-2013 Pre-Screening Prodromal - RBD clarifications Pre-Screening Genetic Cohort - clarified Assessments/tests clarified, including addition of consent (or withdrawal of consent, if applicable) for future contact about future studies and PD family history data collection for Genetic cohort subjects as selected visits.

Amendment 6 - 29-May-2013 Genetics Coordination Core is added to study. The GCC included Genetic Cohort PD Subjects, Genetic Cohort Unaffected Subjects and Genetic Registry Subjects.

Amendment 5 - 27-Nov-2012 Olfactory and RBD subjects added as the Prodromal cohort.

Amendment 4 - 30-Mar-2012 Addition of 18F-AV-133 VMAT-2 PET Imaging for participating U.S. sites and Australia. (Refer to 18F-AV-133-PPMI companion protocol).

Number of sites increased from 21 to 24. Addition of cognitive categorization and diagnostic features assessments.

Amendment 3 - 15-Jul-2011 Addition of SWEDD subjects to study design. Blood Sampling Advisement to collect research samples in a fasted state.

Amendment 2 - 19-May-2011 Changed visit window from 30 days to 45 days for Baseline visit to be completed.

Section on DAT and SPECT Imaging - section changed to account for subject travel to the Institute for Neurodegenerative Disorders to conduct SPECT scanning and injection of either DaTSCAN or BCIT.

Main Protocol - PPMI will be a five-year natural history study (a minimum of 3-year involvement for each subject) of de novo idiopathic PD patients and healthy controls. This study will also include a SWEDD (subjects without evidence of dopaminergic deficit)and Prodromal populations.

All subjects will be comprehensively assessed at baseline and every three to six months thereafter. Subjects will undergo clinical (motor, neuropsychiatric and cognitive) and imaging assessments and will donate blood, urine, and cerebral spinal fluid (CSF). A blood sample for DNA will be collected. Data will be collected by each site under uniformly established protocols and data will be analyzed and stored at designated core facilities.

ELIGIBILITY:
Inclusion Criteria:

Parkinson Disease (PD) Subjects:

* A diagnosis of Parkinson disease for 2 years or less at Screening.
* Confirmation from imaging core that screening DAT scan is consistent with dopamine transporter deficit, or if applicable a VMAT-2 PET scan consistent with vesicular monoamine transporter deficit.
* Not expected to require PD medication with at least 6 months from Baseline.
* Male or female age 30 years or older at time of PD diagnosis.

Healthy Control (HC) Subjects:

• Male or female age 30 years or older at Screening.

Exclusion Criteria:

Parkinson Disease (PD) Subjects:

* Currently taking levodopa, dopamine agonists, MAO-B inhibitors, amantadine or other PD medication.
* Has taken levodopa, dopamine agonists, MAO-B inhibitors or amantadine within 60 days of Baseline.
* Has taken levodopa or dopamine agonists prior to Baseline for more than a total of 60 days.
* Received any of the following drugs that might interfere with DAT imaging: Neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative, within 6 months of Screening.
* Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.

If applicable, currently taking medications that are known to cause QT-prolongation, or are currently taking tetrabenazine (TBZ or amphetamine type medications.

* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Use of investigational drugs within 60 days prior to Baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).

Healthy Control (HC) Subjects:

* Current or active neurological disorder.
* First degree relative with idiopathic PD (parent, sibling, child).
* MoCA score < 26.
* Received any of the following drugs that might interfere with DAT imaging: Neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative, within 6 months of Screening.

If applicable, currently taking medications that are known to cause QT-prolongation, or are currently taking tetrabenazine (TBZ) or amphetamine type medications.

* Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Use of other investigational drugs within 60 days prior to baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).

SWEDD Subjects:

All PD criteria apply, as above, except a SWEDD subject must have confirmation from imaging core that screening dopamine transporter SPECT scan shows no evidence of dopamine transporter deficit or if applicable a VMAT-2 PET scan shows no evidence of vesicular monoamine transporter deficit.

Prodromal Subjects:

Inclusion Criteria (Prodromal Subjects) 4.2.7.1. Subjects must have at least one of the following characteristics:

Hyposmia:

1. Male or female age 60 years or older
2. Confirmation from olfactory core that olfaction as determined by UPSIT is at or below the 10th percentile by age and gender

REM Behavior Disorder (RBD):

1. Male or female age 60 years or older
2. Confirmation from sleep core that subject's Polysomnography (PSG) meets criteria for RBD

LRRK2:

1. Male or female age 60 years or older
2. Written confirmation or documentation from testing facility that the individual is LRRK2 mutation positive 4.2.7.2. Confirmation from imaging core that screening dopamine transporter SPECT scan is read as eligible (see below). About 80 subjects will have a range of DAT deficit similar to subjects with early PD (mild to moderate DAT deficit). About 20 subjects will be selected with no DAT deficit or minimal DAT deficit similar in age, gender, and risk profile to those with mild to moderate DAT deficit. 4.2.7.3. Ability to provide written informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations. 4.2.7.4. Willing and able to comply with scheduled visits, required study procedures and laboratory tests. 4.2.7.5. Women may not be pregnant, lactating or planning pregnancy during the course of the study. Includes a negative urine pregnancy test on day of screening scan prior to injection (DaTSCAN).

Exclusion Criteria (Prodromal Subjects)

1. Current or active clinically significant neurological disorder or psychiatric disorder (in the opinion of the Investigator).
2. GDS score greater than or equal to 10 (GDS score of 5 - 9 requires Investigator discretion to enter study).
3. STAI Form Y-1 greater than or equal to 54 requires Investigator discretion to enter study.
4. A clinical diagnosis of dementia63 as determined by the investigator (Appendix 1).
5. A clinical diagnosis of Parkinson disease at the Screening visit as determined by the Investigator.
6. Received any of the following drugs that might interfere with dopamine transporter SPECT imaging: Neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative, within 6 months of Screening.
7. Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
8. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
9. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
10. Use of investigational drugs or devices within 60 days prior to Baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).
11. Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).

Genetic Cohort: Parkinson Disease Subjects - Inclusion:

1. Patients must have at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting remor or bradykinesia) or either asymmetric resting tremor or asymmetric bradykinesia.
2. A diagnosis of Parkinson Disease for 7 years or less at screening.
3. Hoehn and Yahr state <4 at baseline
4. Male or female age 18 years or older
5. Willingness to undergo genetic testing and to be informed of genetic testing results.
6. Confirmation of mutation in LRRK2, GBA or SNCA
7. For subjects taking any drugs that might interfere with dopamine transporter SPECT imaging (Neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine or amphetamine derivative must be willing and able from a medical standpoint to hold the medication for at least 5 half-lives prior to screening DatSCAN(TM) imaging.

Exclusion:

1. Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
2. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis or clinically significant coagulopathy or thrombocytopenia.

Genetic cohort - Unaffected Individuals

Inclusion:

1. Male or female age 45 years or older at baseline with LRRK2 or GBA mutation and/or first degree relative with a LRRK2 or GBA mutation or
2. Male or female age 30 years or older at baseline with a SNCA mutation and/or a first degree relative with a SNCA mutation.
3. Unaffected subjects at high risk of LRRK2, GBA or SNCA mutation due to first degree relative with a LRRK2, GBA or SNCA mutation may choose either to be informed of the results or remain unaware of the results.
4. Unaffected subjects from an ethnic or geographic group knkown to have relatively high risk of LRRK2, GBA or SNCA mutation such as people of Ashkenazi Jewish or Basques descent) and who have a family member (either alive or deceased) who has/had PD must be willing to be informed of their own testing results.
5. Willingness to undergo genetic testing
6. For subjects taking any of the following drugs that might interfere with dopamine transporter SPECT imaging (neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine or amphetamine derivative) must be willing and able from a medical standpoint to hold the medication for at least 5 half-lives prior to DatSCAN imaging.

Exclusion:

1. A clinical diagnosis of PD
2. Current treatment with anticoagulants (e.g. coumadin, heparin) that might preclude safe completion of the lumbar puncture.
3. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis or clinically significant coagulopathy or thrombocytopenia.

Genetic Registry - Inclusion:

1. Individual with a LRRK2, GBA or SNCA mutation and/or a first degree relative with a LRRK2, GBA or SNCA mutation.
2. Male or female age 18 years or older
3. Willingness to undergo genetic testing, but may choose either to be informed of the results or remain unaware of the results.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mean Rates of Change | Baseline to 156 months
  The mean rates of change and the variability around the mean of clinical, imaging and biomic outcomes in early PD patients, and where appropriate the comparison of these rates between PD patient subsets and between various subsets (including, but not limited to: PD vs. healthy subjects, PD vs. SWEDD, PD vs. prodromal, PD with and without LRRK2, GBA or SNCA mutation, unaffected LRRK2, GBA or SNCA mutation carriers vs. healthy controls) at study intervals ranging from 3 months to 36 months. Specific examples of outcomes include MDS-UPDRS, dopamine transporter imaging striatal uptake, vesicular monoamine transporter type-2 uptake, and serum and CSF alpha-synuclein. PD patient subsets may be defined by baseline assessments, genetic mutations, progression milestones and/or rate of clinical, imaging, or biomic change.

SECONDARY OUTCOMES:
Comparison between Rates of Change | Study intervals ranging from 3 months to 156 months
  Comparison between the rates of change in the mean of clinical, imaging and biomic outcomes in various subsets (including, but not limited to: early PD vs. healthy subjects, PD vs. SWEDD, PD vs. prodromal, PD with and without LRRK2, GBA or SNCA mutation, unaffected LRRK2, GBA or SNCA mutation vs. healthy controls)
Prevalence of measures of clinical, imaging and biomic outcomes in various subsets ( | study intervals ranging from baseline to 156 months.
  Including, but not limited to: early PD patients, healthy subjects, PD vs SWEDDs, PD vs prodromal, PD with and without LRRK2, GBA or SNCA mutation, unaffected LRRK2, GBA or SNCA mutation carriers vs. healthy subjects.
Predictive Value | Baseline to 156 months
  To establish the predictive value of early clinical non-motor features, baseline imaging and biomic outcomes for future course of disease.
To examine the proportion of SWEDD subjects that have a change in their clinical management at 24 months | Baseline to 156 Months
  SWEDD Clinical Diagnosis and Management Questionnaire.
Exploratory Analysis | Baseline to 156 months
  Exploratory analysis to estimate the percentage of Prodromal subjects with one or more risk characteristics [hyposmia (<10th percentile for age and gender), RBD, or LRRK2, GBA or SNCA genetic mutation, and baseline DaTSCAN binding showing minimal to moderate DAT deficit] that phenoconvert to PD within 2 years, and an exploratory analysis to examine whether the baseline DaTSCAN binding or progression of clinical, imaging, or biospecimen markers may predict those subjects likely to phenoconvert.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Marek, MD, Study Chair — Institute for Neurodegenerative Disorders; John Q. Trojanowski, MD, PhD, Study Director — University of Pennsylvania; Arthur W. Toga, PhD, Study Director — University of California, Los Angeles; Tatiana Froud, PhD, Study Director — Indiana University; Karl Kieburtz, MD, Study Director — Clinical Trials Coordination Center; Andrew Singleton, PhD, Study Director — Laboratory of Neurogenetics; National Institute on Aging NIH; John P Seibyl, MD, Study Director — Institute for Neurodegenerative Disorders; Christopher Coffey, PhD, Study Director — Clinical Trials Statistical and Data Management Center, University of Iowa
Locations (34):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Research Institute, Sun City, Arizona
  - University of California San Diego, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - The Parkinson's Institute, Sunnyvale, California
  - Institute For Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease& Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Beth Israel Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati/Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health &Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Univ of Washington and VA Puget Sound Health Care System, Seattle, Washington
- Macquarie University, Sydney, Australia
- Innsbruck Medical University, Innsbruck, Austria
- Hospital Pitie-Salpetriere, Paris, France
- Germany (2):
  - Paracelsus-Elena Klinik, Kassel
  - University of Tuebingen, Tübingen
- Foundation for Biomedical Research of the Academy of Athens, Athens, Greece
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Universita Federico II, Napoli
  - University of Salerno, Salerno
- St. Olavs Hospital, Trondheim, Norway
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
- Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Tsukita K, Kikuya A, Yoshimura K, Nakanishi E, Matsumoto R, Takahashi R. Temporal Dynamics and Cross-Sectional and Longitudinal Factors Associated With Motor Reserve and Outcome in Patients With Parkinson Disease. Neurology. 2026 Jan 27;106(2):e214475. doi: 10.1212/WNL.0000000000214475. Epub 2025 Dec 26. PMID 41453126
- [Derived] Liu Y, Chen M, Chen P, Lin X, Chen S, Liu C, Wang D, Deng H, Li Q, Wu Y. Machine learning-based stratification of mild cognitive impairment in Parkinson's disease: a multicenter cross-sectional analysis. BMC Med Inform Decis Mak. 2025 Oct 15;25(1):384. doi: 10.1186/s12911-025-03215-0. PMID 41094519
- [Derived] Tuena C, Repetto C, Ibanez A, Magni G, Stramba-Badiale M, Riva G. Embodied concepts in Parkinson's disease: Insights from fruits versus animals semantic fluency impairments. Neuropsychology. 2025 Oct;39(7):610-618. doi: 10.1037/neu0001026. Epub 2025 Jul 24. PMID 40705614
- [Derived] Pisani S, Gosse L, Aarsland D, Ray Chaudhuri K, Ballard C, Ffytche D, Velayudhan L, Bhattacharyya S. Parkinson's disease psychosis associated with accelerated multidomain cognitive decline. BMJ Ment Health. 2024 Jul 23;27(1):1-10. doi: 10.1136/bmjment-2024-301062. PMID 39043465
- [Derived] Park M, Lee YG. Association of Family History and Polygenic Risk Score With Longitudinal Prognosis in Parkinson Disease. Neurol Genet. 2023 Dec 8;10(1):e200115. doi: 10.1212/NXG.0000000000200115. eCollection 2024 Feb. PMID 38169864
- [Derived] Tsukita K, Sakamaki-Tsukita H, Kaiser S, Zhang L, Messa M, Serrano-Fernandez P, Takahashi R. High-Throughput CSF Proteomics and Machine Learning to Identify Proteomic Signatures for Parkinson Disease Development and Progression. Neurology. 2023 Oct 3;101(14):e1434-e1447. doi: 10.1212/WNL.0000000000207725. Epub 2023 Aug 16. PMID 37586882
- [Derived] Wang C, Zhou C, Guo T, Jiaerken Y, Yang S, Xu X, Hu L, Huang P, Xu X, Zhang M. Current coffee consumption is associated with decreased striatal dopamine transporter availability in Parkinson's disease patients and healthy controls. BMC Med. 2023 Jul 25;21(1):272. doi: 10.1186/s12916-023-02994-5. PMID 37491235
- [Derived] Kim R, Kang N, Byun K, Park K, Jun JS. Prognostic significance of peripheral neutrophils and lymphocytes in early untreated Parkinson's disease: an 8-year follow-up study. J Neurol Neurosurg Psychiatry. 2023 Dec;94(12):1040-1046. doi: 10.1136/jnnp-2022-330394. Epub 2023 Jul 14. PMID 37451695
- [Derived] Weintraub D, Picillo M, Cho HR, Caspell-Garcia C, Blauwendraat C, Brown EG, Chahine LM, Coffey CS, Dobkin RD, Foroud T, Galasko D, Kieburtz K, Marek K, Merchant K, Mollenhauer B, Poston KL, Simuni T, Siderowf A, Singleton A, Seibyl J, Tanner CM; Parkinson's Progression Markers Initiative. Impact of the Dopamine System on Long-Term Cognitive Impairment in Parkinson Disease: An Exploratory Study. Mov Disord Clin Pract. 2023 Apr 25;10(6):943-955. doi: 10.1002/mdc3.13751. eCollection 2023 Jun. PMID 37332638
- [Derived] Brumm MC, Pierz KA, Lafontant DE, Caspell-Garcia C, Coffey CS, Siderowf A, Marek K. Updated Percentiles for the University of Pennsylvania Smell Identification Test in Adults 50 Years of Age and Older. Neurology. 2023 Apr 18;100(16):e1691-e1701. doi: 10.1212/WNL.0000000000207077. Epub 2023 Feb 27. PMID 36849448
- [Derived] Kim R, Park S, Yoo D, Jun JS, Jeon B. Association of Physical Activity and APOE Genotype With Longitudinal Cognitive Change in Early Parkinson Disease. Neurology. 2021 May 11;96(19):e2429-e2437. doi: 10.1212/WNL.0000000000011852. Epub 2021 Mar 31. PMID 33790041
- [Derived] Simuni T, Brumm MC, Uribe L, Caspell-Garcia C, Coffey CS, Siderowf A, Alcalay RN, Trojanowski JQ, Shaw LM, Seibyl J, Singleton A, Toga AW, Galasko D, Foroud T, Nudelman K, Tosun-Turgut D, Poston K, Weintraub D, Mollenhauer B, Tanner CM, Kieburtz K, Chahine LM, Reimer A, Hutten S, Bressman S, Marek K; Parkinson's Progression Markers Initiative Investigators. Clinical and Dopamine Transporter Imaging Characteristics of Leucine Rich Repeat Kinase 2 (LRRK2) and Glucosylceramidase Beta (GBA) Parkinson's Disease Participants in the Parkinson's Progression Markers Initiative: A Cross-Sectional Study. Mov Disord. 2020 May;35(5):833-844. doi: 10.1002/mds.27989. Epub 2020 Feb 19. PMID 32073681
- [Derived] Simuni T, Uribe L, Cho HR, Caspell-Garcia C, Coffey CS, Siderowf A, Trojanowski JQ, Shaw LM, Seibyl J, Singleton A, Toga AW, Galasko D, Foroud T, Tosun D, Poston K, Weintraub D, Mollenhauer B, Tanner CM, Kieburtz K, Chahine LM, Reimer A, Hutten SJ, Bressman S, Marek K; PPMI Investigators. Clinical and dopamine transporter imaging characteristics of non-manifest LRRK2 and GBA mutation carriers in the Parkinson's Progression Markers Initiative (PPMI): a cross-sectional study. Lancet Neurol. 2020 Jan;19(1):71-80. doi: 10.1016/S1474-4422(19)30319-9. Epub 2019 Oct 31. PMID 31678032
- [Derived] Simuni T, Caspell-Garcia C, Coffey CS, Weintraub D, Mollenhauer B, Lasch S, Tanner CM, Jennings D, Kieburtz K, Chahine LM, Marek K. Baseline prevalence and longitudinal evolution of non-motor symptoms in early Parkinson's disease: the PPMI cohort. J Neurol Neurosurg Psychiatry. 2018 Jan;89(1):78-88. doi: 10.1136/jnnp-2017-316213. Epub 2017 Oct 6. PMID 28986467
- [Derived] Latourelle JC, Beste MT, Hadzi TC, Miller RE, Oppenheim JN, Valko MP, Wuest DM, Church BW, Khalil IG, Hayete B, Venuto CS. Large-scale identification of clinical and genetic predictors of motor progression in patients with newly diagnosed Parkinson's disease: a longitudinal cohort study and validation. Lancet Neurol. 2017 Nov;16(11):908-916. doi: 10.1016/S1474-4422(17)30328-9. Epub 2017 Sep 25. PMID 28958801
- [Derived] Smith KM, Xie SX, Weintraub D. Incident impulse control disorder symptoms and dopamine transporter imaging in Parkinson disease. J Neurol Neurosurg Psychiatry. 2016 Aug;87(8):864-70. doi: 10.1136/jnnp-2015-311827. Epub 2015 Nov 3. PMID 26534930
- [Derived] Oliveira FP, Castelo-Branco M. Computer-aided diagnosis of Parkinson's disease based on [(123)I]FP-CIT SPECT binding potential images, using the voxels-as-features approach and support vector machines. J Neural Eng. 2015 Apr;12(2):026008. doi: 10.1088/1741-2560/12/2/026008. Epub 2015 Feb 24. PMID 25710187